CLINICAL TRIAL: NCT00314782
Title: A Phase I Study of ZD4054 (Zibotentan) in Combination With Docetaxel in 2 Parts, an Open-Label, Non-Randomized, Dose-Finding Part and a Double-Blind, Placebo-Controlled, Randomized Dose Expansion Part, in Patients With Metastatic Hormone-Refractory Prostate Cancer
Brief Title: Phase I Study of ZD4054 (Zibotentan) and Docetaxel in Patients With Metastatic HRPC
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D4320C00020; 4054IL/0020
Record Dates: First submitted 2006-04-13; First posted 2006-04-17 (Estimated); Last update posted 2013-03-12 (Estimated); Status verified 2010-03

CONDITIONS: Prostate Cancer
Keywords: metastatic hormone-refractory prostate cancer (HRPC)
MeSH Terms: conditions — Prostatic Neoplasms | interventions — ZD4054; Docetaxel

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (4):
- Part A (Experimental): Part A (dose-finding): ZD4054 (Zibotentan) 10 mg oral tablet once daily, with docetaxel 75mg/m^2 intravenous infusion once per cycle
  Interventions: Drug: ZD4054 (Zibotentan); Drug: Docetaxel
- Part A (ZD4054 (Zibotentan) 15 mg + docetaxel) (Experimental): Part A (dose-finding): ZD4054 (Zibotentan) 15 mg oral tablet once daily, with docetaxel 75mg/m^2 intravenous infusion once per cycle
  Interventions: Drug: ZD4054 (Zibotentan); Drug: Docetaxel
- Part B (Experimental): Part B (randomised, placebo-controlled): ZD4054 (Zibotentan) Maximum Tolerated Dose (MTD), 15mg, oral tablet once daily, with docetaxel 75mg/m^2 intravenous infusion once per cycle
  Interventions: Drug: ZD4054 (Zibotentan); Drug: Docetaxel
- Part B (placebo) (Experimental): Part B (randomised, placebo-controlled): Matching placebo oral tablet once daily, with docetaxel 75mg/m^2 intravenous infusion once per cycle
  Interventions: Drug: Docetaxel; Drug: Placebo

INTERVENTIONS:
Drug: ZD4054 (Zibotentan) — oral tablet
  Other Names: Zibotentan
  Arms: Part A; Part A (ZD4054 (Zibotentan) 15 mg + docetaxel); Part B
Drug: Docetaxel — intravenous infusion
  Other Names: Taxotere®
Drug: Placebo
  Arms: Part B (placebo)

SUMMARY:
Two-part, multi-center study design to establish a maximum tolerated dose (MTD) of ZD4054 in combination with docetaxel and to explore its safety, tolerability, pharmacokinetic (PK) profiles and clinical efficacy in patients with metastatic hormone-refractory prostate cancer (HRPC)

ELIGIBILITY:
Inclusion Criteria:

* Provision of informed consent
* Histological or cytological confirmation of prostate cancer
* Evidence of metastatic disease on CT scan, MRI, or bone scan
* Surgically or continuously medically castrated with LHRH analogue
* Progressive disease after most recent therapy

  * Disease progression by CT/MRI
  * Bone scan progression: appearance of 1 or more new lesions since last bone scan
  * Rising PSA
* World health organization (WHO) performance status 0 to 2
* Life expectancy of 12 weeks or longer

Exclusion Criteria:

* Use of anti-hormonal therapies (including ketoconazole, aminoglutethimide, finasteride and anti-androgen therapies) within 4 weeks of starting study treatment, except for bicalutamide and nilutamide which are excluded within 6 weeks of starting study treatment. Estramustine or estrogens, if taken, have to be stopped at least 4 weeks before starting treatment.
* Definite or suspected personal history or family history of adverse drug reactions, or hypersensitivity to drugs that are endothelin antagonist; history of severe hypersensitivity reactions to drugs formulated with polysorbate 80.
* Prior cytotoxic chemotherapy for metastatic prostate cancer
* Radiotherapy within 4 weeks before the start of study therapy
* Systemic radionuclide therapy (ie strontium chloride Sr89, 186Re-labeled HEDP, or 153Sm-EDTMP pentasodium) within 12 weeks before entering study
* Use of potent CYP450 inhibitors (such as itraconazole, ritonavir, indinavir, erythromycin, troleandomycin, clarithromycin, diltiazem, verapamil) within 2 weeks before study entry.
* Use of potent CYP450 inducers (such as phenytoin, rifampicin, carbamazepine and phenobarbitone, St. John's Wort) within 2 weeks before study entry.

NOTE: Dexamethasone is a known inducer of CYP2D6 and CYP3A4 but is not considered exclusionary for purposes of this study.

* New neurologic symptoms or signs consistent with acute or evolving spinal cord compression confirmed by magnetic resonance imaging (MRI) (except for those previously treated and have stable symptoms).
* History of past or current epilepsy, epilepsy syndrome, or other seizure disorder
* History of Migraine or chronic headache
* Symptomatic central nervous system (CNS) metastases
* Absolute Neutrophil Count (ANC) <1.5 x 109/L (1,5000/mm3)
* Platelet count < 100 x 109/L (100,000/mm3)
* Serum bilirubin greater than the upper limit of normal (ULN)
* Alanine amino transferase (ALT) or aspartate amino transferase (AST) greater than 1.5 times the upper limit of normal (ULN)
* Creatinine clearance <50 mL/min
* QT interval corrected for heart rate by the Barrett Formula (QTc) > 470 msec at screening
* New York Heart Association (NYHA) class II-IV Heart Disease
* Myocardial infarction (heart attack) within past 3 months
* CTCAE grade ≥2 Peripheral Neuropathy
* Treatment with a non-approved or investigational drug within 30 days before study entry
* Evidence of any other significant clinical symptoms, abnormal laboratory findings or recent surgery that patients has not recovered from that make it undesirable for the patient to participate in the study in the opinion of the investigator(s)
* Involvement in the planning and conduct of the study
* Previous treatment in the present study

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2006-03; Primary Completion 2008-03 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
Part A: Maximum Tolerated Dose (MTD) | Part A: Cycle 1 ('Primary analysis' corresponding to data cut-off 5th March 2008)

CONTACTS AND LOCATIONS:
Overall Officials: AstraZeneca Emerging Oncology Medical Science Director, MD, Study Director — AstraZeneca
Locations (9):
- United States (3):
  - Research Site, Buffalo, New York
  - Research Site, Greenville, South Carolina
  - Research Site, Nashville, Tennessee
- Germany (3):
  - Research Site, Berlin
  - Research Site, Dresden
  - Research Site, Rostock
- United Kingdom (3):
  - Research Site, London
  - Research Site, Plymouth
  - Research Site, Surrey